CLINICAL TRIAL: NCT05394311
Title: Developing & Testing the Feasibility of a Sports-based Mental Health Promotion Intervention for Adolescents in Nepal: a Community Engagement Approach
Brief Title: Testing the Feasibility of a Sports-based Mental Health Promotion Intervention for Adolescents in Nepal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Transcultural Psychosocial Organization Nepal (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MR/T040181/1
Record Dates: First submitted 2022-05-09; First posted 2022-05-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Wellness

STUDY DESIGN:
Intervention Model Description: A parallel-group, two-arm, superiority, cluster-randomised controlled trial with 1:1 allocation to intervention and control arms will be used in the study. Two cross-sectional household surveys of adolescents, one at baseline and one at end line will be conducted.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm - sport based mental health promotion program (Experimental): The experimental arm will receive an intervention for around 10 months' period after baseline data collection.
  Interventions: Other: sports based mental health promotion program
- Control group - treatment as usual (No Intervention): This group receive the intervention available in the existing health care and education system in the study area.

INTERVENTIONS:
Other: sports based mental health promotion program — sports related programs
  Other Names: sports related program
  Arms: Intervention arm - sport based mental health promotion program

SUMMARY:
Each year, one in five adolescents experiences a mental disorder like depression or anxiety, and the rate is rising. Depression is a common mental disorder, one of the leading global causes of Disability Adjusted Life Years among adolescents, and can lead to learning, behavioural and social impairment, as well as comorbid cardiovascular disease and mental illness in adulthood. An intervention is needed that can protect adolescents from mental disorders, is accessible to all adolescents, and is cheap and easy to sustain. One such intervention is mental health promotion, which focuses on improving positive behaviors and characteristics that protect mental health. There is already a strong evidence base for treatment and indicated prevention approaches, but a lack of research on mental health promotion interventions. In low resourced settings like Nepal, interventions need to be short of duration, and be carried out by lay people in the communities to make them sustainable and feasible to implement on a broader scale. The aim of this study is to develop and test the feasibility and acceptability of an intervention that uses sports groups to engage and improve the mental health of adolescents in Nepal.

DETAILED DESCRIPTION:
Depression and anxiety are the leading contributors to the global burden of disease among young people, accounting for over a third (34.8%) of years lived with disability, and contributing significantly to excess mortality through suicide. Adolescence is the peak age of onset for most mental health conditions, with approximately 50% of lifetime mental health conditions having their onset by mid-adolescence. Adolescent depression in turn predicts several adverse life trajectories, such as failure to complete secondary school, unemployment and unplanned pregnancy or parenthood. Early intervention programmes for adolescents can promote mental health, prevent mental disorders, and prevent risky behaviours and other unhealthy lifestyle choices. These programmes have the potential to make positive contributions to adolescents' health, and to their health in later life. One such intervention is mental health promotion, which focuses on improving positive behaviors and characteristics that protect mental health. Mental health promotion is a strategy to improve the positive behaviors and characteristics that protect mental health

A pilot trial will be conducted to assess the feasibility, acceptability and utility of the intervention and trial design; safety and delivery of the intervention in the community settings; and to identify issues around training, supervision and outcomes measures. A household survey will be conducted at baseline and end line data collection points. After a baseline data collection, the implemention of the intervention will be conducted for around 10 months' period, and then collect the follow-up (end line) data with adolescents.

A parallel-group, two-arm, superiority, cluster-randomised controlled trial with 1:1 allocation to intervention and control arms will be done. In total there will be four clusters (2 control and 2 intervention clusters). The unit of randomization will be a geographic village cluster of ~1000 people (approx 160 adolescents in each cluster). Clusters will be separated geographically which will mitigate risk of contamination in the control arm. A researcher will visit each household in the clusters and ask if there are any adolescents living in the household. Where appropriate consent is obtained, the researcher will then interview eligible adolescents using a smartphone or tablet pre-programmed with the survey. The main trial analysis will be a cross-sectional comparison of data from the endline survey, adjusted for baseline differences. Intervention activities will be open to all adolescents aged 12-19 living in the community to participate. The acceptability of the intervention, randomisation, tools, uptake, utility of the intervention, facilitators' fidelity to the manual, mental health outcome trends, and cost of design and delivery of the intervention will be assessed. The intervention process data will be also collected. This will include FGDs and interviews with adolescents and their parents, facilitators and trainers to explore feasibility and acceptability of the intervention and study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Any adolescent boy or girl aged 12-19 years
2. Adolescents in or out of school
3. Married or unmarried
4. Who lives in the study clusters
5. Able to speak and listen

Exclusion Criteria:

1. Participants who are unable to provide a written consent
2. People having severe mental illness or severe physical disability
3. Participants who are planning to move from the study sites during the study period

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 640 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in mental wellbeing of adolescents | From baseline to endline (10 months after the intervention)
  Mental wellbeing is a marker of mental health promotion and defined as subjective evaluation of life satisfaction. This will be measured using the Warwick Edinburgh Mental Wellbeing Scale. The scale is scored by summing responses to each item answered on a 1 to 5 Likert scale where '1' indicates 'none of the time' and '5' indicates 'all of the time'. The minimum scale score is 14 and the maximum is 70 with with higher scores indicating a higher level of mental wellbeing.

SECONDARY OUTCOMES:
Self-efficacy | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Schwarzer General Self-Efficacy (GSE) Scale will be used to measure self-efficacy. For each item there is a four choice response scale where '1' indicates 'not at all true and '4' indicates 'exactly true'. The minimum scale score is 10 and the maximum is 40 with a higher score indicating a higher self-efficacy.
Self-esteem | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Rosenberg Self-Esteem Scale (RSES) will be used to measure self-esteem. RSES is a 10-item scale that measure global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be uni-dimensional. All items are answered using a 4-point rating scale format ranging from strongly agree '4' to strongly disagree '1'. The scale ranges from 0-30, with higher score indicating high self-esteem.
Emotion regulation | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) will be used to measure emotion regulation. It is a 10-item self-report measure consisting of two kinds of emotion regulation strategies, namely, cognitive reappraisal (CR) (6 items) and expressive suppression (ES) (4 items). It has a five points rating scale where '1' indicates 'strongly disagree', and '5' indicates 'strongly agree'. Higher scores on each scale indicate greater use of the corresponding emotional regulation strategy.
Depression | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Depression Self-Rating Scale (DSRS) will be used to measure depression. DSRS has 18-items and the respondents are asked to score their experience of 18 common symptoms of depression in the past one week. It has a 3-point rating scale where '0' indicates 'not at all' and '2' indicates 'always'. The total score of DSRS ranges from 0 to 36 with higher score indicating severity of depression.
Anxiety | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Generalised Anxiety Disorder (GAD-7) will be used to measure anxiety. GAD-7 has 7-items and respondents are asked to score their experience of 7 common symptoms of anxiety in the past two weeks. It has a 4-point rating scale where 0 indicates 'not at all' and 3 indicates 'always'. The minimum scale score is 0 and the maximum is 28 with high score indicating severity of anxiety.
Resilience | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Resilience Scale will be used to measure resilience. RS has 8-items which was adapted from the 25-Item Gail M. Wagnild & Heather M. Young - "The Resilience Scale" (1987) had previously been used in Nepal to determine which items were culturally salient. It has a 4-point rating scale where 0 indicates 'not at all' and 3 indicates 'always'.The total score of RS ranges from 0 to 24 with higher scores indicate higher levels of resilience.
Functional impairment | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Functional impairment scale (FIS) will be used to measure impairment in daily activities. FIS is 10-item scale to assess impairment in daily functioning. It consists of 10-items, representing daily activities that adolescents generally do for themselves, family and community. It has a 4-point rating scale where 0 indicates 'not at all' and 3 indicates 'always'. The total score of FIS ranges from 0 to 30 with higher score indicating more impairment in daily activities.
Pro-social behaviour | Baseline (T0) before start of the intervention and Endline (T1) 10-month after baseline
  Strengths and Difficulties Questionnaire (SDQ) will be used to measure prosocial behavior. SDQ is a 25-items scale which assesses emotional symptoms, conduct problems, hyperactivity-inattention, peer relationship problems, and prosocial behaviors of adolescent. Prosocial sub-scale of SDQ assesses the social behavior of adolescents. It has three choice response scales 'not true, 'somewhat true' and 'certainly true'. The total score of SDQ prosocial behavious sub-scale ranges from 0 to 10 with higher score indicating more engagement in social behavious.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Gautam, MD, Study Director — Transcultural Psychosocial Organization Nepal
Locations (1):
- Patharisanischare municiaplity and Kanepokhari rural municipality, Biratnagar, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose-Clarke K, Rimal D, Morrison J, Pradhan I, Hodsoll J, Jaoude GA, Moore B, Banham L, Richards J, Jordans M, Prost A, Lamichhane N, Regmee J, Gautam K, Luitel NP. Development and testing the feasibility of a sports-based mental health promotion intervention in Nepal: a protocol for a pilot cluster-randomised controlled trial. Pilot Feasibility Stud. 2023 Aug 24;9(1):149. doi: 10.1186/s40814-023-01324-z. PMID 37620929